CLINICAL TRIAL: NCT07085975
Title: The Safety, Feasibility, and Repeatability of Inhaled ATP Cough Challenges
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: McMaster University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ATP-17839
Record Dates: First submitted 2025-07-17; First posted 2025-07-25 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Chronic Cough (CC); Asthma
Keywords: adenosine triphosphate; chronic cough; asthma; cough hypersensitivity syndrome
MeSH Terms: conditions — Chronic Cough; Asthma; cough hypersensitivity syndrome | interventions — Adenosine Triphosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Adenosine 5'triphosphate (Experimental)
  Interventions: Drug: Adenosine 5'-triphosphate

INTERVENTIONS:
Drug: Adenosine 5'-triphosphate — Participants will inhale increasing doubling concentrations of adenosine 5'-triphosphate dissolved in 0.9% saline through the Aerogen Solo vibrating mesh nebulizer.

SUMMARY:
The inhalation of adenosine 5'-triphosphate (ATP) to evoke cough (ATP cough challenge) is becoming increasingly used as a tool to measure cough hypersensitivity in patients with chronic cough. However, the safety, feasibility, and repeatability of this procedure is not widely known. In this study, we will perform ATP cough challenges in healthy individuals and in patients with mild asthma and chronic cough to better understand the safety, feasibility, and repeatability of these challenges. Such information will guide the future conduct of ATP cough challenges to measure cough hypersensitivity and identify patients who may better respond to ATP-blocking therapies.

ELIGIBILITY:
Phase 1: Healthy individuals

Inclusion Criteria:

Eligible participants in Phase 1 will include healthy adults (≥18 years old) with:

1. Normal spirometry; and
2. No current or past medical history of chronic cough or other respiratory diseases.

Exclusion Criteria:

We will exclude healthy individuals meeting the following:

(1) Are a current or former smoker with a >5 pack-year history and abstinence ≤6 months;

1. Unable to perform acceptable and reproducible spirometry;
2. Have unresolved symptoms of upper respiratory tract infection within 6 weeks prior to the first study visit;
3. Have had a lower respiratory tract infection or pneumonia within 6 weeks prior to the first study visit;
4. Presence of other primary pulmonary disorders, including pulmonary embolism, pulmonary hypertension, lung cancer, cystic fibrosis, radiologically-proven emphysema, severe bronchiectasis, or severe interstitial lung disease; or
5. History of psychiatric illness, drug, or alcohol abuse that could interfere with participation in the study.
6. History of clinically-significant cardiovascular disease, including coronary artery disease, aortic aneurysm, or stroke in the last 3 months;
7. Those with serious medical conditions or those who are not on stable medication(s) for their condition(s);
8. Those with immune system disorders, severe allergy, or on allergy-specific immunotherapy;
9. Any other condition, that, in the opinion of the qualified investigator, may adversely affect the participant's ability to complete the study or its measures or pose significant risk to the participant;
10. Pregnant or breastfeeding;
11. Women of child-bearing potential who:

    1. Do not agree to use a medically approved method of birth control for the duration of the study. All hormonal birth control must have been in use for a minimum of 3 months. Acceptable methods of birth control include oral contraceptives, hormone birth control patch, vaginal contraceptive ring, injectable contraceptives, or hormone implant, double-barrier method, intrauterine devices, non-heterosexual lifestyle or agrees to use contraception if planning on changing to heterosexual partner(s), vasectomy of partner at least 6 months prior to screening. Females who are not of child-bearing potential will be defined as females who have undergone a sterilization procedure (e.g., hysterectomy, bilateral oophorectomy, bilateral tubal ligation, complete endometrial ablation) or have been post-menopausal for at least 1 year prior to screening.

Phase 2: Patients with RCC/UCC and mild-steroid naïve asthma

Inclusion Criteria:

Eligible participants will include adults (≥18 years old) with:

1. RCC/UCC for >1 year, demonstrated by a normal chest radiograph and no airflow obstruction (FEV1/FVC>0.7/LLN) with either:

   1. Insufficient improvement in cough despite treatment targeting any underlying condition(s) contributing to the cough (RCC); or
   2. Cough for which an underlying cause has not been determined despite thorough investigation (UCC).
2. Mild steroid-naïve asthma who demonstrate evidence of a positive screening methacholine (PC20<16 mg/mL); symptoms of cough, shortness of breath, chest tightness, and wheeze, that, in the opinion of the qualified investigator, are well-controlled; and those have not used inhaled or oral corticosteroids for the past month.

Exclusion Criteria:

Cohort-specific exclusion criteria include the following:

For the RCC/UCC cohort:

(1) Current smoker or ex-smoker with ≥20 pack-year history and abstinence ≤6 months;

For the mild steroid-naïve asthma cohort:

1. Current smoker or ex-smoker with ≥20 pack-year history and abstinence ≤6 months;
2. History or exacerbation or uncontrolled symptoms within the last month prior to the first study visit; and
3. Use of inhaled or oral corticosteroids within the last month prior to the first study visit.

We will exclude participants meeting any of the following criteria from the study:

1. Unable to perform acceptable and reproducible spirometry;
2. Unresolved symptoms of upper respiratory tract infection within 6 weeks prior to the first study visit;
3. Lower respiratory tract infection or pneumonia within 6 weeks prior to the first study visit;
4. Presence of other primary pulmonary disorders, including pulmonary embolism, pulmonary hypertension, lung cancer, cystic fibrosis, radiologically-proven emphysema, severe bronchiectasis, or severe interstitial lung disease;
5. History of psychiatric illness, drug, or alcohol abuse that could interfere with participation in the study;
6. History of clinically-significant cardiovascular disease, including coronary artery disease, aortic aneurysm, or stroke in the last 3 months;
7. Those with serious medical conditions or those who are not on stable medication(s) for their condition(s);
8. Those with immune system disorders, severe allergy, or on allergy-specific immunotherapy;
9. Any other condition, that, in the opinion of the qualified investigator, may adversely affect the participant's ability to complete the study or its measures or pose significant risk to the participant;
10. Pregnant or breastfeeding;
11. Female participants of child-bearing potential who:

    1. Do not agree to use a medically approved method of birth control for the duration of the study;
    2. Have not been using hormonal birth control for a minimum of 3 months prior to screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2025-08-05 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
The mean %FEV1 change from baseline at incremental doses of ATP | Until the end of the ATP cough challenge
Symptoms of wheeze measured on the mBorg scale at incremental doses of ATP | Until the end of the ATP cough challenge
Symptoms of chest tightness measured on the mBorg scale at incremental doses of ATP | Until the end of the ATP cough challenge
Symptoms of shortness of breath measured on the mBorg scale at incremental doses of ATP | Until the end of the ATP cough challenge
The mean change in oxygen saturations (SpO2) from baseline at incremental doses of ATP | Until the end of the ATP cough challenge
The intra-class correlation of measures obtained from repeat ATP cough challenges | Baseline to 1 week
The frequency of adverse events | Baseline to 1 week
Total maximum number of evoked coughs (Emax) by any dose of ATP | Until the end of the ATP cough challenge
The dose of ATP that induces at least 50% of the maximal cough response (ED50) | Until the end of the ATP cough challenge
The dose of ATP that induces at least 5 coughs (C5) | Until the end of the ATP cough challenge
The dose of ATP that induces at least 2 coughs (C2) | Until the end of the ATP cough challenge

CONTACTS AND LOCATIONS:
Locations (1):
- Respiratory Research Lab, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided